CLINICAL TRIAL: NCT04417764
Title: Safety and Effect Assessment of TACE in Combination With Autologous PD-1 Knockout Engineered T Cells by Percutaneous Infusion in the Paitents With Advanced Hepatocellular Carcinoma.
Brief Title: TACE Combined With PD-1 Knockout Engineered T Cell in Advanced Hepatocellular Carcinoma.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Wei Wang,MD, Principal for The Institute for Cell Transplantation and Gene Therapy, Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CellTransplant&GeneTherapy2020
Record Dates: First submitted 2020-05-29; First posted 2020-06-05 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: CRISPR Cas 9; TACE; PD-1 knockout engineered T cells; Advanced hepatocellular carcinoma; Locally administered treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combined PD-1 knockout T cell treatment (Experimental)
  Interventions: Procedure: Transcatheter arterial chemoembolization; Biological: PD-1 knockout engineered T cells

INTERVENTIONS:
Procedure: Transcatheter arterial chemoembolization — The patients are plan to operated by Transcatheter arterial chemoembolization(TACE).
Biological: PD-1 knockout engineered T cells — The PD-1 knockout engineered T cells are prepared from autologous origin using CRISPR Cas9 technology. The patients are plan to receive 3 or more cycles of PD-1 knockout engineered T cells infusion by percutaneous fine needle liver puncture with a 4-weeks interval. A total of 1 to 3× 10^9 PD-1 edited T cells will be infused each cycle. Patients continued receiving treatment unless they had unacceptable adverse effects, or progressive disease confirmed by CT or they withdrew consent.

SUMMARY:
This study will evaluate the safety and effect of transcatheter arterial chemoembolization (TACE)combined with percutaneous transhepatic PD-1 knockout engineered T cell infusion in the Paitents with advanced hepatocellular carcinoma(HCC). Blood and tissue samples will also be collected for research purposes.

DETAILED DESCRIPTION:
This is a clinical study to investigate the safety and effect of transcatheter arterial chemoembolization (TACE) in combination with PD-1 knockout engineered T cells in the Paitents with advanced hepatocellular carcinoma. TACE would block the blood supply of the tumor to achieve ischemic, hypoxic andnecrotic effects. The PD-1 knockout engineered T cells were also prepared from autologous origin using CRISPR Cas9 technology. The patients performed one TACE treatment followed by 3 cycles of PD-1 edited T cells by percutaneous infusion in the peripheral of tumor under the guide of CT every four weeks. The safety and clinical efficacy will be evaluated. biomarkers and immunological markers will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable hepatocellular carcinoma;
2. More than 18 years old;
3. Patients diagnosed with hepatocellular carcinoma by histopathology or imagings;
4. Liver function ChildPugh ≤7 points, Physical strength score ECOG-pts 0-1 points;
5. Maximum tumor diameter ≤10cm, tumor number ≤10, no vascular invasion or extrahepatic metastasis;
6. Other organs of the whole body function well;
7. Sign the informed consent;
8. Passed the review by the ethics committee.

Exclusion Criteria:

1. Less than 18 or more than 70 years old;
2. Lack of autonomous decision-making ability;
3. ECOG score >2, cachexia or multiple organ failure;
4. Metastases; The tumor was diffuse or metastasized widely and the expected survival time was less than 3 months.
5. Uncorrectable coagulation dysfunction with a history of bleeding; Organ transplant;
6. Patients with severe autoimmune diseases; Iodine contrast agent allergy; High allergic constitution;
7. The main portal vein was completely blocked by cancer embolism, with little collateral vascular formation;
8. Severe infection; AIDS, syphilis infection;
9. T cell lymphoma;
10. Patients with mental illness, severe trauma or other stress conditions;
11. Pregnant or nursing women;
12. Abnormal peripheral blood routine detection;
13. Failing to comply with the study protocol to complete the diagnosis and treatment project; Failed ethics committee review.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | up to 2 years
  Number of participants with Adverse Events using Common Terminology Criteria for Adverse Events (CTCAE v4.03) in patients.

SECONDARY OUTCOMES:
Response Rate | up to 12 months
  To evaluate the objective response rate (ORR) ,refers to the proportion of patients whose tumors shrink to a certain extent and remain unchanged for a certain period of time, including patients with CR+PR.Tumors are assessed at baseline, the 8th week, the 16th week,the 24th week, and once every 12 weeks during the treatment and follow-up period per RECIST1.1.
Time to First Response | up to 2 years
  To evaluate time to first response, defined as the time from the first cell infusion to the first observed complete response (CR) or partial response (PR).
Duration of Response | up to 2 years
  To evaluate the duration of response (DOR), defined as the time from the first observed CR or PR to the first observed PD or death from any cause.
Progression Free Survival | up to 2 years
  To evaluate the progression free survival (PFS), defined as the time from the first cell infusion to the first observed PD or death from any cause.
Overall Survival | up to 2 years
  To evaluate the overall survival (OS), defined as the time from the first cell infusion to death.

CONTACTS AND LOCATIONS:
Locations (1):
- The 3rd Xiangya Hospital of Central South University, Changsha, Hunan, China